CLINICAL TRIAL: NCT05179941
Title: Pilot Feasibility Study of Dynamic Contrast-enhanced Fluorescence Imaging to Guide Total Shoulder Arthroplasty Approach
Brief Title: Subscapularis Indocyanine Green Perfusion Pilot Study
Acronym: ICG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Responsible Party: Principal Investigator, John-Erik Bell, Orthopaedics staff physician, Dartmouth-Hitchcock Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: STUDY02001327
Record Dates: First submitted 2021-12-17; First posted 2022-01-06 (Actual); Last update posted 2023-08-04 (Actual); Status verified 2023-08

CONDITIONS: Shoulder Pain; Shoulder Arthritis; Shoulder Arthroplasty
Keywords: Orthopaedic; Shoulder; Joint Replacement; ICG; Indocyanine green
MeSH Terms: conditions — Shoulder Pain | interventions — Perfusion; Indocyanine Green

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- patients requiring a shoulder arthroplasty (Experimental): Patients will be administered Food and Drug Administration (FDA) approved Indocyanine green (ICG) through intravenous injection and imaged by a FDA approved surgical fluorescence imaging device. Both ICG fluorescence and the imaging system have been used for routine clinical practice for many years. ICG fluorescence imaging utilizes intravenously injected ICG, which is a fluorescent dye that is FDA approved for clinical use, illuminated with near-infrared light. The ICG dye is indirectly activated and the dynamic fluorescence due to meniscal perfusion can be captured by an FDA approved imaging system.
  Interventions: Procedure: Perfusion with Indocyanine green

INTERVENTIONS:
Procedure: Perfusion with Indocyanine green — Infusion of Indocyanine green to determine perfusion of the subscapularis tendon change after tenotomy vs peel technique and subsequent intra-operative repair.

SUMMARY:
The Purpose of this pilot study is to evaluate the feasibility of open wide-field imaging of indocyanine green ingress and egress during total shoulder arthroplasty. This study also hopes to characterize the relationship between tissue perfusion measured with DCE-FI and different approaches and techniques used in total shoulder arthroplasty. The long term goal of this study is to determine if there is a potential relationship between perfusion and patient reported outcomes and subscapularis failure.

DETAILED DESCRIPTION:
Shoulder arthroplasty is a commonly utilized and routinely successful surgery performed for management of glenohumeral joint arthritis. Upwards of 90% of primary anatomic total shoulder arthroplasty surgeries are considered successful. Albeit rare, complications do occur. Complications include glenoid or humeral component loosening, periprosthetic fracture, infection and rotator cuff failure. Of the four muscles that comprise the rotator cuff, the subscapularis is of particular concern in total shoulder arthroplasty surgery due to the approach used to access the glenohumeral joint. The deltopectoral approach is the standard approach used for shoulder arthroplasty and necessitates performing a subscapularis takedown in order to obtain adequate visualization of the glenohumeral joint. Three techniques to perform a subscapularis takedown are common, with an absence of consensus in the literature as to which technique is superior. The techniques include a subscapularis peel, and a subscapularis tenotomy.

Each subscapularis takedown technique requires repair at the conclusion of the procedure when performing shoulder arthroplasty. Repair is crucial for proper force coupling of the shoulder to keep the humeral head implant centered on the glenoid component. Takedown is still performed in a reverse total shoulder arthroplasty but repair is not required to maintain stability. Each takedown technique is reliant on a tendon to tendon interface for healing. Failure of the subscapularis tendon repair can result in pain, instability, decreased functional outcomes and ultimately the need for revision surgery. Subscapularis tendon failure can sometimes be asymptomatic, however it can also be symptomatic and present with the aforementioned signs. Subscapularis failure rates may approach 50% in long term studies although symptomatic cases likely occur in less than 1% of total shoulder arthroplasties . Due to the devastating impact on patients with symptomatic subscapularis failure, there is interest in investigating which subscapularis takedown technique produces the best outcomes. Prior randomized controlled trials as well as systematic reviews have previously been conducted looking at these different takedown techniques, but demonstrated no statistically significant difference in primary endpoints of subscapularis strength at various time endpoint and no statistically significant difference in patient reported outcomes. These prior studies did not evaluate subscapularis perfusion post repair, adequate perfusion is necessary for healing to occur with any subscapularis takedown technique.

The takedown method of the subscapularis has previously been shown to have no statistically significant differences with regards to strength, or patient reported outcomes, however if there was a difference noted in tendon perfusion post repair this may provide rationale to choose one technique over another as improved perfusion may correlate to lower risk of repair failure.

The data acquired using the SPY Elite or SPY PHI or EleVision will be deanonymized and exported to a secure PC for additional analysis and processing. The analysis techniques will be more sophisticated than the current commercial system, and involve a correction for the patient-specific arterial input function (AIF) -the cardiac and circulatory variations that can modify the time and manner in which the ICG dye arrives in the imaging field-of-view.

Indocyanine green (ICG) is a well-studied water soluble, light absorbing tracer that has been used in other capacities to help quantify tissue perfusion during surgery. ICG is able to be injected into a patient intravenously and subsequently circulate systemically while bound to albumin, quickly undergoing hepatic metabolism in just several minutes. The concentration of ICG in specific tissue is able to be quantified as a surrogate for tissue perfusion. ICG due to its IV administration and quick metabolism is able to help quantify perfusion in real time, such as intra-operatively. Systemic reviews as well as case studies, most commonly in plastic surgery, have been performed showing its utility to determine adequate or inadequate perfusion in downstream tissue in situations where microanastomoses are performed, such as with flaps and in hand surgery. Other studies have also been conducted showing the ability to use ICG as a surrogate for tissue perfusion in the achilles paratenon in humans and in rabbits who had undergone rotator cuff repair to determine tissue perfusion after different types of repair. The use of ICG imaging in orthopaedic surgery is relatively nascent, and our institution as well as other collaborators have demonstrated its promise in these applications.

ELIGIBILITY:
Inclusion criteria:

* - Participant must be 18 years of age or older
* - Meet clinical and radiographic parameters necessary to undergo shoulder arthroplasty
* - Subscapularis tendon intact clinically on exam or via advanced imaging
* - Subject has the ability to have their shoulder arthroplasty completed using either the tenotomy or peel technique.

Exclusion criteria:

* - Inability of patient to provide informed consent
* - Iodine allergy
* - Subscapularis tendon tear or concern for tear
* - Incarceration
* - Pregnant women
* - Patients less than 18 years of age
* - Prior deltopectoral approach to the ipsilateral shoulder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2022-02-11 (Actual); Primary Completion 2022-12-13 (Actual); Study Completion 2022-12-13 (Actual)

PRIMARY OUTCOMES:
measurement of change to tendon blood supply during total shoulder arthroplasty | Baseline, up to 2 hours
  The primary study outcome is to evaluate the ingress and egress in tendon and tissue blood flow in patients undergoing a total shoulder repair.

SECONDARY OUTCOMES:
measurement of change to tendon blood supply using different techniques used in total shoulder arthroplasty | Baseline, up to 2 hours
  To characterize the relationship between tissue perfusion with different approaches used in total shoulder arthroplasty

CONTACTS AND LOCATIONS:
Overall Officials: John-Erik Bell, MD, Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (1):
- Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire, United States

DOCUMENTS (1):
  • Study Protocol (2021-12-29): https://cdn.clinicaltrials.gov/large-docs/41/NCT05179941/Prot_000.pdf